CLINICAL TRIAL: NCT06086600
Title: Comparison of Instrument Assisted Soft Tissue Mobilization Versus Dynamic Oscillatory Stretch Technique in Females Wearing High Heels
Brief Title: Instrument Assisted Soft Tissue Mobilization Versus Dynamic Oscillatory Stretch Technique in Females Wearing High Heels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01610
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Behavior, Social
Keywords: instrument assisted soft tissue mobilization; dynamic oscillatory stretch technique; high heel users
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument Assisted Soft Tissue Mobilization (Experimental): Graston tool on gastrocnemius and soleus muscle. Conventional treatment will include
  * Hot pack for 10-15 min (calf muscles)
  * Stretching exercises of gastro-soleus (10reps x 2Sets).
  * Post session : Cold pack for 5 minutes (calf muscles)
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Dynamic oscillatory stretch technique (Active Comparator): Dynamic oscillatory stretch technique on gastrocnemius and soleus muscle10reps x2 second hold oscillation x 3 sets.
  Conventional treatment will include
  * Hot pack for 10-15 min (calf muscles)
  * Stretching exercises of gastro-soleus (10reps x 2 Sets).
  * Post session : Cold pack for 5 minutes (calf Muscles
  Interventions: Other: Dynamic oscillatory stretch technique

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — give gentle strokes from proximal to distal to check for trigger point or taut band. After knowing the exact location, give gentle strokes with minimal pressure in all directions by keeping the instrument in 30 to 60 degree angle. Application time will be between 40- 120 seconds.
  Conventional treatment will include
  * Hot pack for 10-15 min (calf muscles)
  * Stretching exercises of gastro-soleus (10reps x 2Sets).
  * Post session : Cold pack for 5 minutes (calf muscles)
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Dynamic oscillatory stretch technique — Passively dorsiflexe the ankle to a point of the first stretch sensation. The next component to DOS, 2- second, passive stretch with slow oscillations at end range was applied. This procedure is repeated 10 times in each set with total of 3 sets .Therefore,10reps x2 second hold oscillation x 3 sets are given.Conventional treatment will include
  * Hot pack for 10-15 min (calf muscles)
  * Stretching exercises of gastro-soleus (10reps x 2Sets).
  * Post session : Cold pack for 5 minutes (calf muscles
  Arms: Dynamic oscillatory stretch technique

SUMMARY:
Rationale of this research is to compare the effect of instrument assisted soft tissue mobilization and dynamic oscillatory stretch technique on gastro soleus muscles flexibility with shortened calf muscle-tendon unit (MTU),thicker and stiffer Achilles tendon in individual wearing high heel. This study will observe effect in all range of motion of ankle joint. In Pakistan no previous research is conducted, that compare the effect of IASTM and DOST in females wearing high heel.

DETAILED DESCRIPTION:
Regular wearing of high heels would lead to shortening of the fascicles of the gastrocnemius muscle together with changes in the mechanical properties of the Achilles' Tendon, by the continuous ankle plantar flexion cause by the heel lift resulting in functional alteration. The purpose of the study is to identify the optimal technique for alleviating the symptoms in patients with high heel syndrome. It is a randomized controlled trial.Sample size is total 54 participants which would be divided into two groups, 27 each.Non-probability Convenience Sampling will be used and participants are randomly assigned into GROUP A(IASTM) and GROUP B (DOST) through sealed envelope methods after baseline assessment. All participants in both groups were evaluated on two occasions: (i) baseline (ii) at 12th session.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* Duration of wearing heels: minimum 1 year
* Wearing heels for minimum 3 times a week and 5 hours a day.
* Heel height: 2" and above
* Ankle Dorsiflexion ROM: decreased dorsiflexion (about 17 degrees)
* Pain scale showing more than 3.

Exclusion Criteria:

* DVT
* Musculoskeletal injury or surgery of lower limb.
* Acute Cardio-Respiratory or Neurological condition.
* Medical or surgical co-morbidities

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Ankle Range of Motion | 4th week
  Goniometer is used to measure ankle dorsiflexion, Plantarflexion, inversion, eversion ROM and it is use to assess and monitor patient's mobility to track progress during rehabilitation.
Lower Extremity Functional Scale (LEFS) | 4th week
  The Lower Extremity Functional Scale (LEFS) is a commonly used tool in physical therapy and rehabilitation to assess the functional abilities of patients with lower extremity impairments. It is a self-reported questionnaire that consists of 20 items, each with five response options ranging from 0 (unable to perform) to 4 (able to perform without difficulty). The scores on the LEFS range from 0 to 80, with higher scores indicating better function.
NUMERIC PAIN RATING SCALE | 4th week
  The numeric pain rating scale is used to measure pain intensity. It typically ranges from 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain. Patients are asked to rate their pain on this scale, with the healthcare provider using the rating to help guide treatment decisions. It is a simple and effective way to communicate pain intensity, and can be useful in tracking changes in pain over time.

SECONDARY OUTCOMES:
ROM ankle dorsi flexion | 4th week
  changes from baseline to final session
ROM ankle plantar flexion | 4th week
  changes from baseline to final session
ROM ankle inversion | 4th week
  changes from baseline to final session
ROM ankle eversion | 4th week
  changes from baseline to final session

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Gulberg green campus of Riphah International University, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien HL, Lu TW, Liu MW. Effects of long-term wearing of high-heeled shoes on the control of the body's center of mass motion in relation to the center of pressure during walking. Gait Posture. 2014 Apr;39(4):1045-50. doi: 10.1016/j.gaitpost.2014.01.007. Epub 2014 Jan 19. PMID 24508016
- [Background] Pannell SL. The postural and biomechanical effects of high heel shoes: a literature review. Journal of Vascular Surgery. 2012.